CLINICAL TRIAL: NCT05268198
Title: A Phase 1, Randomized, Blinded, Placebo-Controlled, First-in-Human, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of APR002 Administered by Inhalation in Healthy Volunteers
Brief Title: SAD Study of APR002 Investigating the Safety/Tolerability, Pharmacokinetics/Pharmacodynamics in Healthy Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Global Health Drug Discovery Institute (Other)
Collaborators: CMAX Clinical Research Pty Limited (Unknown); Avance Clinical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: APR002-NEB-001
Record Dates: First submitted 2022-02-17; First posted 2022-03-07 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — APR002; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention/Treatment (Experimental): Single dose, oral inhalation (nebuliser solution)
  Interventions: Drug: APR002
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APR002 — Active Investigational Product
  Other Names: TLR7 agonist
  Arms: Intervention/Treatment
Drug: Placebo — Placebo
  Other Names: 0.9% Sodium Chloride; Saline
  Arms: Placebo

SUMMARY:
This study will investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of single ascending doses of APR002 in healthy subjects.

DETAILED DESCRIPTION:
A Phase 1, Randomized, Blinded, Placebo-Controlled, First-in-Human, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of APR002 Administered by Inhalation in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women aged 18 to 55 years (inclusive) with suitable veins for cannulation or repeated venipuncture.
* Women can be of childbearing potential and must have been stable on a highly effective contraceptive method for at least 3 months prior to Visit 1 (screening) and be willing to continue on the chosen contraceptive method
* Male subjects should be willing to use a condom (with spermicide) to prevent pregnancy and drug exposure of a female partner and refrain from donating sperm or fathering a child from the day of the investigational product administration until 3 months
* Have a body mass index (BMI) between 18 and 32 kg/m2 and weigh at least 45 kg.

Exclusion Criteria:

* History or presence of clinically significant medical (e.g., chronic obstructive pulmonary disease, asthma, COVID-19, etc.) or psychiatric condition or disease
* Abnormal vital signs, after minutes rest, defined as any of the following (SBP > 140 mmHg, Diastolic blood pressure (DBP) > 90 mmHg, Heart rate < 40 or > 99 beats per minute)
* Prolonged QTcF > 450 ms or family history of long QT syndrome

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of APR002 in healthy subjects as assessed by incidence of treatment-emergent adverse events according to CTCAE v5.0 criteria | Screening up to Day 14
  Safety assessments will include evaluation of incidence of treatment-emergent adverse events (AEs) according to CTCAE v5.0 criteria, including vital signs, resting electrocardiogram (ECG) parameters, standard hematology, chemistry, urinalysis and other tests

SECONDARY OUTCOMES:
Pharmacokinetics of APR002 in healthy subjects as assessed by maximum plasma concentration (Cmax) towards determination of the optimal pharmacokinetic dose | Day 1 to Day 3
  Determination of maximum plasma concentration (Cmax)
Pharmacokinetics of APR002 in healthy subjects as assessed by time to maximum concentration (Tmax) towards determination of the optimal pharmacokinetic dose | Day 1 to Day 3
  Determination of time to maximum concentration
Pharmacokinetics of APR002 in healthy subjects as assessed by plasma exposure (AUC0-t, AUC0-inf) determination of the optimal pharmacokinetic dose | Day 1 to Day 3
  Determination of plasma exposure (AUC0-t, AUC0-inf)
Pharmacokinetics of APR002 in healthy subjects as assessed by terminal elimination half life (t1/2) determination of the optimal pharmacokinetic dose | Day 1 to Day 3
  Determination of terminal half life
Pharmacokinetics of APR002 in healthy subjects as assessed by apparent volume of distribution during the terminal elimination phase after inhalation (extravascular) administration for determination of the optimal pharmacokinetic dose | Day 1 to Day 3
  Determination of volume of distribution (CL/F and Vz/F)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Weitzman, Study Director — Global Health Drug Discovery Institute
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia